CLINICAL TRIAL: NCT04237454
Title: Thermal Imaging Compared to Skeletal Survey for Diagnosis of Fractures in Suspected Inflicted Injury in Children Below 2 Years of Age: A Prospective Diagnostic Accuracy Study
Brief Title: Thermal Imaging Compared to Skeletal Survey in Children Below 2 Years
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Children's NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SCH-13-067f
Record Dates: First submitted 2020-01-03; First posted 2020-01-23 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Fracture; Abuse Physical
MeSH Terms: conditions — Fractures, Bone

STUDY DESIGN:
Intervention Model Description: Thermal Imaging
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Infrared Imaging undertaken (Experimental)
  Interventions: Device: Thermal Imaging Camera

INTERVENTIONS:
Device: Thermal Imaging Camera — To develop a non-ionising radiation-based method of excluding fractures in children with suspected physical abuse

SUMMARY:
When a child less than 2 years old attends the Emergency Department (ED) with an injury, carers should offer an explanation. When there is no explanation or if the explanation is inconsistent & because the child cannot say what happened, the doctor will need to consider all possible causes including child abuse. To help exclude abuse, the doctor will request x-rays of all the child's bones to make sure there are no other unexplained fractures. This requires up to 20 x-rays, which are called a skeletal survey. Even if there are no fractures, some or all of the x-rays will be repeated in the following 7-21 days, because by that time any fractures will have started to heal and so are easier to see than on the first skeletal survey. It means that if a doctor is worried about abuse, the child may need to have up to 40 x-rays, which amounts to a significant radiation dose (more than 6 months of natural UK background radiation) & increases the child's lifetime risk of getting cancer. 79 to 97 out of 100 skeletal surveys performed are normal. While it is of paramount importance to identify if a child is being abused, it is also important to minimise radiation dose. A camera which detects light and heat given off by the body has shown promise in some areas of medical practice. We plan to compare the results from the camera to those of the skeletal survey in 40 children below 2 years of age attending our hospital over a 6-month period. We hope to demonstrate that this technology can be used to further select children who should have a skeletal survey, reducing radiation dose in children without missing those who are being abused and sending them home to be abused again.

ELIGIBILITY:
Inclusion Criteria:

* Children between 1 month and 2 years of age having initial/follow-up skeletal survey for investigation of suspected abuse
* Healthy Control children

Exclusion Criteria:

* 1. Informed consent withheld by main carer/guardian for the skeletal survey (court order would then be issues) 2. Informed consent for participation in the research study withheld 2. Situations where informed consent cannot be obtained (e.g. inability of carer/guardian to understand written English) 3. Postmortem cases (inclusion of the demised would unduly complicate the consent process for this small pilot study)

Ages: 1 Month to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2017-04-11 (Actual); Study Completion 2017-04-11 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of thermal imaging for fracture detection compared to skeletal survey as the gold standard | 6 months
  Diagnostic accuracy (sensitivity, specificity, positive and negative predictive value) of thermal imaging compared to the full skeletal survey as gold standard

SECONDARY OUTCOMES:
Potential radiation dose reduction - calculated on the basis of known radiation exposure of the images that form the skeletal survey | 6 months
  Radiation dose saving of a protocol that only images those areas of abnormality seen on thermal imaging compared to the full skeletal survey as gold standard
Carer acceptability/preference of the imaging modalities | 6 months
  Descriptive statistics based on responses to a non-validated questionnaire on carer experiences of both imaging techniques

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Research Facility, Sheffield, South Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No